CLINICAL TRIAL: NCT01086995
Title: Weaning And Variability Evaluation
Brief Title: Weaning And Variability Evaluation (WAVE)
Acronym: WAVE
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: OH2007-588
Record Dates: First submitted 2010-03-12; First posted 2010-03-15 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Extubation
Keywords: extubation; weaning; mechanical ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine if variability in heart and breathing rates can be used to predict successful weaning. We are collecting data to determine whether or not subtle differences in heart rate and respiratory function will help physicians to decide if a patient is ready to be weaned.

DETAILED DESCRIPTION:
In this prospective observational pilot study, mechanically ventilated patients weaning or near extubation (i.e. within 1-5 days) were selected to undergo continuous heart rate (EKG waveform at 500 Hz) and respiratory rate (expired CO2 waveform at 100 Hz) recording. The data was collected as per standard practice by the bedside monitor (Phillips Intelivue MP70). A portable CPU with TrendfaceTM software was used to download the data for variability analysis. All decisions on timing of SBTs and extubation were left to the discretion of the treating team who were unaware of the variability results. SBT's were repeated daily from trial onset until extubation patient permitting.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been requiring mechanical ventilation for >48 hours.
* At least partial reversal of the condition precipitating invasive ventilation.
* Stabilization of "other" organ system failures (i.e. no worsening).
* The patient is able to tolerate pressure support ventilation ≤14 cm H2O (SpO2 ≥ 90% with FiO2 ≤ 40% and PEEP ≤ 10 cm H2O)
* The patient is hemodynamically stable (off vasopressors or on low levels of vasopressors).
* Stable neurological status (no deterioration in the last 24 hors, intact respiratory drive and ICP < 20).
* The patient has intact airway reflexes (adequate cough with suctioning and a gag reflex).

Exclusion Criteria:

* Allergy to skin adhesives or a contraindication to placing electrocardiogram adhesives (e.g. severe psoriasis).
* Do not reintubate order documented on chart or anticipated withdrawal of life support.
* Tracheostomy
* Known or suspected severe myopathy or neuropathy (i.e. myasthenia gravis, Guillain-Barré syndrome) or quadriplegia.
* Severe heart failure or Grade IV left ventricular function.
* Prior extubation during ICU stay.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated patients weaning or near extubation (i.e. within 1-5 days) in the intensive care unit.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2007-11; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Continuous heart rate and respiratory rate waveforms | at time of sponataneous breathing trial (at least 48 hours after intubation and within 24 hours of extubation)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Seely, MD, PhD, FRCSC, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital General Campus, Ottawa, Ontario, Canada